CLINICAL TRIAL: NCT06450301
Title: Is Thin Endometrial Lining Associated with Senescent Endometrial Cells
Brief Title: Senescent Endometrial Cells in Patients with Thin Endometrial Lining
Status: Recruiting | Type: Observational
Sponsor: Trio Fertility (Other)
Responsible Party: Principal Investigator, Dr. Robert F. Casper, Scientific Director, MD, FRCSC, REI, University of Toronto
Other Study IDs: 3533
Record Dates: First submitted 2024-05-28; First posted 2024-06-10 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Asherman's Syndrome; Thin Endometrial Lining; Cell Senescence
MeSH Terms: conditions — Gynatresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will measure the percentage of senescent cells in endometrial biopsies by Sudan Black-B (SBB) immunohistochemistry, since this is a specific marker of cell senescence and can be performed on formalin fixed, paraffin-embedded tissue. This assay also allows us to test archived samples for women in the control group who have already had an endometrial biopsy. We will also freeze part of the endometrial biopsy sample for RNA extraction for senescent biomarker expression (BMI-1, p16lnka4, p14ARF, Cyclin-D1, and CDK4 by RT-PCR) and protein determination (western blotting) for confirmation of the SBB staining results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Thin endometrial lining: Patients following long-term use of oral contraceptives with known thin endometrial lining (less than 7mm, confirmed in at least two cycles and unresponsive to estrogen-induced growth).
  We will ask each woman to undergo an endometrial biopsy as part of the study during their luteal phase.
  Interventions: Procedure: Endometrial Biopsy
- Asherman's syndrome: Patients with Asherman's syndrome following Dilation and curettage (D&C). We will ask each woman to undergo an endometrial biopsy as part of the study during their luteal phase.
  Interventions: Procedure: Endometrial Biopsy
- Control: Patients already scheduled to undergo an endometrial biopsy for infertility management.
  We will ask each woman to undergo an endometrial biopsy as part of the study during their luteal phase. In some cases, we may be able to access archived endometrial samples from women in the control group who agree to participate and who have already had an endometrial biopsy.
  Interventions: Procedure: Endometrial Biopsy

INTERVENTIONS:
Procedure: Endometrial Biopsy — An endometrial biopsy is the removal of a small piece of tissue from the endometrium, which is the lining of the uterus. Endometrial biopsies are commonly done to check for the window of implantation, to determine ovulation or for enhancing implantation (procedure called endometrial scratching). For this purpose, we will use a "Pipelle" catheter. This procedure is very common in gynecologic practice and
  generally considered safe. In most of the cases this procedure is indicated for evaluation of irregular vaginal bleeding, vaginal bleeding in post-menopausal women and for infertility related problems (recurrent implantation failures for example).

SUMMARY:
The goal of this observational study is to determine if thin endometrial lining that is unresponsive to estrogen might be associated with the presence of senescent cells in patients following long-term use of oral contraceptives. The main question it aims to answer is:

Are there any senescent cells present in thin endometrial lining?

During the luteal phase of the cycle, participants will will undergo:

* Gynecologic US to measure the endometrial lining thickness and pattern.
* Endometrial biopsy with Pipelle catheter

DETAILED DESCRIPTION:
The investigators hypothesized that senescent cells in the endometrium may be the cause of the failure of thin endometrium to respond to normal growth stimuli such as estrogen.

The outcome that research team anticipate to measure is the percentage of senescent cells in the endometrial biopsies of women with thin endometrium compared to the control group biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-39
* BMI - up to 35
* Thin endometrium after OCP use
* Asherman's syndrome
* Women already undergoing endometrial biopsy for infertility testing (eg. EMMA testing)
* Women with archived endometrial biopsy samples

Exclusion Criteria:

* Women with systemic disease (Rheumatic disease, DM)
* Women with coagulopathies
* Women with active pelvic inflammatory process
* Uterine anomalies
* Pregnant women
* Any hormonal contraception use or IUD

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We intend to recruit 30 patients following long-term use of oral contraceptives with known thin endometrial lining (less than 7mm, confirmed in at least two cycles and unresponsive to estrogen-induced growth). We will also recruit 20 women with Asherman's syndrome following D&C. We will ask each woman to undergo an endometrial biopsy as part of the study. As a control group, we will recruit 50 patients already scheduled to undergo an endometrial biopsy for infertility management (EMMA testing, endometrial scratching for IVF cycles). Endometrial biopsies are standard procedures during infertility investigations. In some cases, we may be able to access archived endometrial samples from women in the control group who agree to participate and who have already had an endometrial biopsy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Senescent cells presence | Through study completion, an average of 3 years.
  Percentage of senescent cells in the endometrial biopsies of women with thin endometrium compared to the control group biopsies.

CONTACTS AND LOCATIONS:
Locations (1):
- Trio Fertility, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided